CLINICAL TRIAL: NCT03573687
Title: The Effect of Protein Timing and Resistance Exercise on Lipolysis and Fat Oxidation in Resistance-Trained Women
Brief Title: Effects of Protein Timing and Resistance Exercise on Fat Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Michael J. Ormsbee, Assistant Professor, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NPRO
Record Dates: First submitted 2017-01-23; First posted 2018-06-29 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Healthy
Keywords: protein; lipolysis; fat oxidation; resistance training; nutrient timing
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Randomized, crossover, double-blind, acute study with two conditions: nighttime PRO consumption (NP) and daytime PRO consumption (DP).
Who Masked: Participant, Investigator
Masking Description: The supplements will be made by a third party person and premixed, taste-matched, and provided in opaque shaker bottles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RT on Fat Metabolism (Experimental): Determine the extent to which a full-body acute RT protocol will affect intra-RT and post-RT SCAAT lipolytic rate, and post-RT whole-body substrate utilization in RT women compared to baseline measures (independent of Aims 2 and 3).
  Interventions: Other: Resistance Exercise Training
- PRO Timing on Fat Metabolism (Experimental): Assess the differences in overnight and next morning SCAAT lipolytic rate and next-morning whole-body substrate utilization compared to baseline between acute NP and DP consumption trials after a RT bout in RT women.
  Interventions: Dietary Supplement: Micellar Casein Protein; Other: Resistance Exercise Training
- PRO Timing on Markers of Fat Metabolism (Experimental): Assess the differences in overnight and next morning metabolic biomarkers of fat metabolism compared to baseline between acute nighttime PRO (NP) consumption versus daytime PRO (DP) consumption trials after a RT bout in RT women.
  Interventions: Dietary Supplement: Micellar Casein Protein; Other: Resistance Exercise Training

INTERVENTIONS:
Dietary Supplement: Micellar Casein Protein — The micellar casein protein supplement (PRO, total protein content: 30 g, 120 kcals; 30 g micellar protein) and non-caloric sensory-matched placebo (PLA, 0kcals) will be specifically formulated by Dymatize® Nutrition FrieslandCampina® and consumed in a randomized order. Participants will consume the daytime supplement 30 minutes after RT and the nighttime supplement about 30 minutes before bedtime. The supplements will be premixed, taste-matched (chocolate), and provided in opaque shaker bottles.
  Arms: PRO Timing on Fat Metabolism; PRO Timing on Markers of Fat Metabolism
Other: Resistance Exercise Training — Resistance exercise training (RT) will target the full body and exercises will be performed using a barbell. Exercises will be performed in the following order: back squat, bench press, Romanian deadlift, bent-over row, shoulder press, and reverse lunges)

SUMMARY:
The extent to which resistance exercise training and protein timing effects localized (belly fat) and systemic (whole body) fat metabolism in resistance-trained women is unknown. Therefore, this study will assess subcutaneous abdominal adipose tissue lipolytic rate and whole body substrate utilization over the course of two trials: 1) consuming casein protein during the day, and 2) consuming casein protein at night, before bed.

DETAILED DESCRIPTION:
Nighttime eating, and specifically eating after dinner, has attracted significant attention in recent years, particularly for the onslaught of media claiming the negative implications on body weight and overall health. Some studies have indeed indicated that chronically eating high-energy, mixed-meals rich in carbohydrates (CHO) and fats at night contributes to weight gain and abdominal obesity. However, research to support these negative claims is scant. Conversely, the practice of nighttime eating of small protein (PRO) snacks has been widely utilized anecdotally in populations such as bodybuilders in an attempt to avoid catabolism of muscle mass during the sleeping hours.

It has been shown that nighttime consumption of small portions (<200 kcals) of PRO elicits beneficial effects on metabolism such as increased next-morning resting metabolic rate (RMR). Likewise, the combination of nighttime PRO consumption and RT improves factors that contribute to fat loss such as elevated muscle mass due to an increase in muscle protein synthesis and energy expenditure. Further, there is emerging research suggesting the benefits of nighttime PRO consumption on fat metabolism (specifically the subcutaneous abdominal adipose tissue [SCAAT]). The SCAAT is of particular interest in metabolism research, as the upper body subcutaneous tissue (i.e. SCAAT) supplies most of the circulating free fatty acids (FFA) during the overnight hours in lean individuals. Therefore, if one can optimize the timing of dietary PRO during a window at which SCAAT is elevated (nighttime), theoretically, mobilization and oxidation of fats could be optimized.

Research regarding nighttime eating, specifically regarding fat metabolism, is in its infancy, and thus, many gaps in the literature require elucidation. First, and certainly most importantly, the limited research studies examining the effects of nighttime PRO consumption have not methodologically matched for timing of PRO intake. Therefore, it is unclear whether any reported benefits of the published nighttime PRO studies were a consequence of the addition of PRO calories or specifically due to the consumption of PRO at night. Thus, in order to make optimal comparisons and conclusions, it is imperative to study the metabolic effects of dietary PRO consumed at night versus other times of day.

Therefore, the purpose of this project is to: 1) determine the effects of RT on post-exercise lipolytic rate in resistance-trained women; and 2) determine the effects of timing of acute protein PRO ingestion (nighttime PRO consumption [NP] and daytime PRO consumption [DP] trials) after a RT bout on SCAAT lipolytic rate, metabolic rate, and serum hormones (glucose, insulin, growth hormone, adiponectin, glycerol) throughout the day, overnight and into the next morning.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Resistance-trained (able to squat 1.0 times their body weight, and bench press 0.75 times body weight, adapted from ACSM Guidelines and piloted in our laboratory)
* Normal weight (BMI = 18.5-25 kg/m2; body fat <33%)
* Normally menstruating (on or off oral contraceptives)
* Females.

Exclusion Criteria:

* Uncontrolled thyroid dysfunction (not on medication)
* Musculoskeletal disorders
* Currently smoke
* Have milk allergies
* Currently take medications or supplements known to affect substrate metabolism.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Lipolysis | 18 hours
  Lipolysis is the way that fat cells mobilize the stored fat to enter into blood circulation. Lipolysis can be measured using a technique called microdialysis. In short, a semi-permeable probe is inserted into the subcutaneous abdominal adipose tissue (SCAAT, or belly fat). Saline combined with a minute amount of ethanol is perfused into the SCAAT, and interstitial fluid is collected out. The concentration of ethanol in the interstitial fluid sample is an indicator of blood flow within the tissue. Glycerol and free fatty acid concentration is measured to indicated rate of fat metabolism (specifically glycerol). The area under the curve for glycerol concentration over time (AUCgly) will be calculated for each of time point. Microdialysis dialysate samples will be measured during the NP and DP trials at fifteen separate time points throughout each visit.

SECONDARY OUTCOMES:
Hormone Concentrations | 18 hours
  Serum samples will be analyzed for the assessment of glucose, insulin, and growth hormone on collections 1, 3, 4, and 5. Serum glycerol will be assessed at 5 time points. Serum catecholamines will be assessed at time points 1, 2 and 3. The timeline for blood collections is as follows:
  1. During microdialysis probe equilibration (~1600 hours);
  2. Half way through the RT protocol (~1800 hours, after the third exercise: Romanian deadlift)
  3. Thirty minutes after daytime supplement (1900 hours);
  4. Thirty minutes after nighttime supplement (2300 hours), and;
  5. The following morning after RMR (0750 hours)
Fat oxidation | 18 hours
  Fat oxidation is when those stored fats enter into the muscle cells and are able to be oxidized to form energy. Fat oxidation will be quantified by measuring resting metabolic rate (RMR, amount of calories burned at rest) and respiratory exchange ratio (RER, measure of whole-body substrate utilization) using a dilution technique and open-circuit indirect calorimetry (ParvoMedics TrueOne 2400 metabolic cart, Sandy, UT). This technique uses a ventilated hood covering the participants' head and torso. Participants will be asked to remain awake, quiet, and as motionless as possible in a semi-recumbent position in a quiet, dark, climate-controlled isolated room (20-23°C). Resting metabolism will be measured on four separate occasions.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Sports Sciences and Medicine, Florida State University, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Allman BR, Morrissey MC, Kim JS, Panton LB, Contreras RJ, Hickner RC, Ormsbee MJ. Lipolysis and Fat Oxidation Are Not Altered with Presleep Compared with Daytime Casein Protein Intake in Resistance-Trained Women. J Nutr. 2020 Jan 1;150(1):47-54. doi: 10.1093/jn/nxz186. PMID 31504693